CLINICAL TRIAL: NCT03130153
Title: Comparison of Topical Analgesic With Saline Rinses in Post Extraction Healing Among Hypertensive and Non-Hypertensive Patients
Brief Title: Topical Analgesic Versus Saline Mouth Rinses in Post Extraction Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3425-Sur-ERC-14
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Tooth Extraction Site Healing
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hypertensives on Aspirin mouthwash (Experimental)
  Interventions: Drug: Aspirin Powder
- non-hypertensives on Aspirin mouthwash (Active Comparator)
  Interventions: Drug: Aspirin Powder
- hypertensives on Saline mouthwash (Active Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Aspirin Powder — Aspirin powder to be dissolved in water and to be used as mouthwash twice daily for 7 days after tooth extraction.
  Other Names: Acetyl salicylic acid
  Arms: hypertensives on Aspirin mouthwash; non-hypertensives on Aspirin mouthwash
Drug: Normal saline — Normal saline to be used as mouthwash twice daily for 7 days after tooth extraction among non-hypertensive subjects.
  Other Names: 0.9% NaCl; Saline
  Arms: hypertensives on Saline mouthwash

SUMMARY:
There is no evidence based guidelines on using saline rinses for post extraction oral care among hypertensives. Similarly, benefit of orally dissolved topical analgesics in addition to orally administered analgesic is questionable.

DETAILED DESCRIPTION:
Objective: To compare the post dental extraction healing among subjects who took simple analgesic tablets dissolved in water versus those who used saline rinses post operatively.

Methods: A study will be done among patients who underwent dental extractions at AKHSP dental clinic, Karachi, Pakistan. Carious, periodontally mobile, traumatized or broken down teeth among 20-70 years old in either gender will be included.

In addition to the routine prescription of antibiotics and oral analgesics, the hypertensive subjects (n=20) will be advised to take dissolved Aspirin tablet as an oral care while non-hypertensive will be divided into two sub groups (n=20 each), advised saline mouth rinses or dissolved Aspirin for 5 days, respectively.

The outcome (healing of the extraction socket) will be evaluated 7 days from the day of extraction on an ordinal scale.

ELIGIBILITY:
Inclusion Criteria:

* Carious, periodontally mobile, traumatized or broken down teeth needing extraction
* Age 20-70 years, both genders

Exclusion Criteria:

* Diabetes
* Osteoporosis, metabolic bone disease etc.
* Radiation therapy or chemotherapy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Healing of the extraction socket | Seven days from the day of extraction
  1. = "healed or healing well"
  2. = "incomplete healing but progressing"
  3. = "poorly healed open margins and readily bleeding"

CONTACTS AND LOCATIONS:
Overall Officials: Farhan R Khan, BDS MS FCPS, Study Director — AKU
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No